CLINICAL TRIAL: NCT05540548
Title: Contribution of the Podiatrist-Posturologist in the Evaluation of the Link Between the Stabilometric Parameters and the Pain Felt in Patients With Chronic Low Back Pain
Acronym: APLOMB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0522; 2022-A00253-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Kinesiophobia; Pain; Posturology; Stabilometry
MeSH Terms: conditions — Kinesiophobia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic low back pain is one of the major causes of disability worldwide. Knowledge about the pathophysiology of low back pain is insufficient, and an accurate diagnosis can only be obtained in 10 to 15% of cases. The absence of a precise diagnosis leads to a therapeutic challenge due to the large number of treatments available, the overall efficacy of which is low to moderate. Therefore, the identification of subgroups of non-specific chronic low back pain patients is essential and will allow the optimization of therapeutic management. A detailed description of the stabilometric parameters associated with the evaluation of pain, kinematic disturbance and the degree of kinesiophobia would allow us to establish specific postural profiles, to propose a relevant clinical model and to improve the accuracy of the diagnosis of people with chronic low back pain. The objectives of this research project are to evaluate the relationship between stabilometric parameters and pain (main objective), lumbar kinematics, kinesiophobia, and quality of life (secondary objectives) in order to propose specific postural profiles in chronic low back pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from low back pain, possibly associated with painful gluteal radiation in the form of mono or bilateral pygalgia (non-radicular) evolving for at least three months (chronic low back pain
* Understanding and being able to express himself in French
* Giving informed, dated and signed consent

Exclusion Criteria:

* Neurosurgical criteria: (i) presence of clinical signs of compression and/or single or multi-root pain (Lumbosciatica with or without deficit signs, intermittent claudication of the cauda equina roots with possible sphincter signs), (ii) history inflammatory arthropathy (ankylosing spondylitis, rheumatoid arthritis), and (iii) history of lumbar spine surgery.
* Radiographic criteria: (i) presence on the lumbar MRI of multi-level discopathy (more than 2 discopathy), (ii) spinal instability confirmed by CT or MRI (degenerative spondylolisthesis or by isthmic lysis).
* Pregnant or breastfeeding women
* Visually impaired patient
* Patient suffering from neurological and/or orthopedic disorders that may affect balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited within the pain unit of the General Hospital of Valenciennes, within the framework of the multidisciplinary consultation of the optimized pain and dedicated to the low back pain patients, where intervene a neurosurgeon algologist and a podiatrist posturologist.
  The selection of patients enrolled in the multidisciplinary pain consultation dedicated to low back pain patients will be reviewed by the Clinical Study Technician (screening) and checked by the principal investigator before the newsletter is sent.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-06-11 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between the average speed of displacement of the center of pressure measured in the open-eyes position and the level of pain felt in patients suffering from chronic low back pain | Baseline

SECONDARY OUTCOMES:
Correlation between the other stabilometric parameters (mean surface, mean frontal and sagittal position) of postural stability measured in the open-eyes position and the level of pain felt. | Baseline
Correlation between the stabilometric parameters (mean speed, mean surface, mean frontal and sagittal position) of postural stability (measured in the open-eyes position and in the closed-eyes position) and neuropathic pain | Baseline
Correlation of stabilometric parameters (mean speed, mean surface, mean frontal and sagittal position) of postural stability (measured in open-eyes and closed-eyes position) with the degree of kinesiophobia and quality of life. | Baseline
Reproducibility of the stabilometric measurements (average speed, average surface, average frontal and sagittal position) in each of the conditions (in the open-eyes position and in the closed-eyes position). | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VISEUX, Principal Investigator — University Hospital, Lille
Locations (1):
- Service de neurologie CH de Valenciennes, Valenciennes, France